CLINICAL TRIAL: NCT04829318
Title: Open-label Long-Term Extension Study for Participants With Treatment-Resistant Major Depressive Disorder Who Are Continuing Esketamine Nasal Spray Treatment From Study 54135419TRD3013
Brief Title: A Long-Term Extension Study for Participants With Treatment-resistant Major Depressive Disorder Who Are Continuing Esketamine Nasal Spray Treatment
Acronym: ESCAPE-LTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108992; 2020-004291-18 (EudraCT Number); 54135419TRD4010 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2021-04-01; First posted 2021-04-02 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Depressive Disorder, Major
Keywords: Treatment resistant depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Esketamine (Experimental): Participants who were randomly assigned to the esketamine arm in Study 54135419TRD3013 (NCT04338321), had esketamine nasal spray administered through Week 30 (every 2 weeks dosing) or Week 31 (once weekly dosing), completed the maintenance phase at Week 32 will continue to receive esketamine nasal spray once weekly or every 2 weeks along with serotonin-norepinephrine reuptake inhibitor/selective serotonin reuptake inhibitor (SSRI/SNRI) in this long-term extension (LTE) study. The duration of the study participation is 2 years or when esketamine is commercially available.
  Interventions: Drug: Esketamine; Drug: SSRI/SNRI

INTERVENTIONS:
Drug: Esketamine — Esketamine will be self-administered as nasal spray.
Drug: SSRI/SNRI — Participants will continue to take SSRI/SNRI that is approved for use in depression in their country of participation; off-label use of any SSRI/SNRI is not permitted. The continuing SSRI/SNRI dosage may be optimized throughout the study, at the investigator's discretion and based on the summary of product characteristics (SmPC) (or local equivalent, if applicable). During this LTE study, investigators will be allowed to switch individual participant's SSRI/SNRI for tolerability issues.

SUMMARY:
The primary purpose of this study is to assess the long-term safety and tolerability of esketamine nasal spray in combination with a selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) in participants who have completed 32 weeks of esketamine nasal spray treatment in Study 54135419TRD3013 (NCT04338321).

ELIGIBILITY:
Inclusion Criteria:

* Completed the maintenance phase (Week 32) of Study 54135419TRD3013 (NCT04338321) and had esketamine nasal spray in combination with continuing selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI) administered through Week 30 (every 2 week dosing) or Week 31 (once weekly dosing) of Study 54135419TRD3013, and continues to be willing to be treated with esketamine nasal spray
* Must, in the opinion of the investigator, be benefiting from continuation of esketamine nasal spray in combination with their current SSRI/SNRI based on efficacy and tolerability assessed on Day 1 of this study
* Must be medically stable based on the investigator's judgment
* A woman of childbearing potential must have a negative urine pregnancy test on Day 1
* Male participants who are sexually active with a woman of childbearing potential must agree to the following during the intervention period and for at least 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study intervention (that is, esketamine nasal spray), must fulfill the following criteria: must be practicing a highly effective method of contraception with his female partner, must use a condom if his partner is pregnant, and must agree not to donate sperm

Exclusion Criteria:

* Has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Completed Study 54135419TRD3013 while presenting adverse events deemed clinically relevant by the investigator, and which may interfere with safety and well-being of the participant
* Has developed during participation in Study 54135419TRD3013 any of the following cardiovascular-related conditions where an increase in blood pressure or intracranial pressure poses a serious risk: cerebrovascular disease following stroke or transient ischemic attack, aneurysmal vascular disease (including intracranial, thoracic, or abdominal aorta, or peripheral arterial vessels), intracerebral hemorrhage, coronary artery disease following myocardial infarction, unstable angina, or revascularization procedure (example, coronary angioplasty or bypass graft surgery), uncontrolled brady- or tachyarrhythmias that lead to hemodynamic instability, hemodynamically significant valvular heart disease such as mitral regurgitation, aortic stenosis, or aortic regurgitation or heart failure (New York Heart Association [NYHA] Class III-IV) of any etiology
* Significant pulmonary insufficiency, including chronic obstructive pulmonary disease
* Has homicidal ideation or intent, per the investigator's clinical judgment; or has suicidal ideation with some intent to act within 1 month prior to Day 1, per the investigator's clinical judgment; or based on the Columbia-suicide severity rating scale (C-SSRS) performed at Week 32 visit of Study 54135419TRD3013, corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) for suicidal ideation
* Pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 90 days after the last dose of study intervention

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (59):
- Argentina (7):
  - FunDaMos, Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Fundacion Lennox, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Sanatorio Prof Leon S Morra S A, Córdoba
  - Instituto de Neurociencias San Agustin, La Plata
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
- Anima, Alken, Belgium
- Bulgaria (3):
  - Mental Health Center - Rousse, Rousse
  - Multiprofile Hospital for Active Treatment in Neurology and Psychiatry Sveti Naum, Sofia
  - Centre for Mental Health Prof.N.Shipkovenski EOOD, Sofia
- Czechia (7):
  - Psychiatricka ambulance Saint Anne s.r.o., Brno
  - Psychiatricka ambulance, MUDr. Marta Holanova, Brno
  - NeuropsychiatrieHK, s.r.o., Hradec Králové
  - A Shine S R O, Pilsen
  - AD71 s.r.o., Prague
  - Medical Services Prague S R O, Prague
  - Institut Neuropsychiatricke pece, Prague
- Mederon LTD at ARTES, Helsinki, Finland
- Germany (10):
  - Medizinisches Versorgungszentrum LiO GmbH, Berlin
  - Praxis Dr. med. Kirsten Hahn, Berlin
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitätsklinikum Freiburg - Abteilung für Psychiatrie u. Psychotherapie mit Poliklinik, Freiburg im Breisgau
  - Klinische Forschung Hamburg, Hamburg
  - Oberhavel Kliniken GmbH, Hennigsdorf
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Mittweida
  - Danuvius Klinik Pfaffenhofen Fachklinik für Psychiatrie, Psychotherapie und Psychosomatik, Pfaffenhofen
  - Somni Bene GmbH, Schwerin
  - Klinische Forschung Schwerin GmbH, Schwerin
- Greece (3):
  - Psychiatric Clinic 'Agios Charalampos', Heraklion
  - University General Hospital of Rio Patras, Pátrai
  - G Papanikolaou Hospital of Thessaloniki, Thessaloniki
- Hungary (3):
  - Processus Kft, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Petz Aladar Megyei Oktato Korhaz, Győr
- Malaysia (4):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Pengajar Universiti Putra Malaysia, Serdang
  - Hospital Tuanku Jaafar, Seremban
- Poland (9):
  - Mlynowamed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk, Bialystok
  - Osrodek Badan Klinicznych CLINSANTE S C, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Centrum Medyczne Care Clinic Katowice, Katowice
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Specjalistyczny Psychiatryczny Zespol Opieki Zdrowotnej w Lodzi Szpital im. J. Babinskiego, Lodz
  - SPZOZ CSK UM w Lodzi Klinika Zaburzen Afektywnych i Psychotycznych, Lodz
  - Osrodek Badan Klinicznych CLINSANTE S C, Torun
- South Africa (2):
  - Cape Town Clinical Research Centre, Cape Town
  - Gert Bosch Pretoria South Africa, Pretoria
- South Korea (2):
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (3):
  - Hacettepe University Medical Faculty, Ankara
  - Erenkoy Mental Health Hospital, Istanbul
  - Liv Hospital, Samsun

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 183 participants who completed the maintenance phase (Week 32) of study 54135419TRD3013 (NCT04338321) were enrolled and treated in this study.
Groups:
- Esketamine Nasal Spray + Oral Antidepressant (AD): Participants (who received esketamine nasal spray in study 54135419TRD3013 [NCT04338321] through Week 30 [every 2 weeks dosing] or Week 31 [once weekly dosing], and completed the maintenance phase at Week 32), received flexible dose of esketamine nasal spray 28 milligrams (mg) (one spray to each nostril at 0 minute), 56 mg (one spray to each nostril at 0 and 5 minutes) or 84 mg (one spray to each nostril at 0, 5 and 10 minutes) once weekly or every 2 weeks from Day 1 (Week 32 visit of study 54135419TRD3013 until week 104 along with oral AD, serotonin-norepinephrine reuptake inhibitor/selective serotonin reuptake inhibitor (SSRI/SNRI) in this long-term extension (LTE) study. Time 0 minute signified time of first esketamine nasal spray administration to 1 nostril. Esketamine nasal devices contained a total of 28 mg esketamine per device (2 sprays). Only one device was used at a timepoint.
Period: Overall Study
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Started | 183
Treated With Esketamine 28 mg | 2
Treated With Esketamine 56 mg | 68
Treated With Esketamine 84 mg | 113
Treated With Oral AD | 182
Completed | 148
Not Completed | 35
Not completed — Adverse Event | 6
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 19
Not completed — Site terminated by sponsor | 1
Not completed — Sponsor decision | 5
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.07)
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 174
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants analyzed included participants who reported ethnicity.
  Participants
    number analyzed (Participants) | 72
    Hispanic or Latino | 12
    Not Hispanic or Latino | 60
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Participants analyzed included participants who reported race.
  Participants
    number analyzed (Participants) | 72
    American Indian or Alaska Native | 0
    Asian | 6
    Native Hawaiian or Other Pacific Islander | 66
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0
Body mass index [Count of Participants; unit: Participants] — Population: Participants analyzed included participants who reported body mass index in kilograms per meter square (kg/m^2).
  Participants
    Underweight <18.5 kg/m^2: number analyzed (Participants) | 155
    Underweight <18.5 kg/m^2 | 5
    Normal 18.5 to <25 kg/m^2: number analyzed (Participants) | 155
    Normal 18.5 to <25 kg/m^2 | 63
    Overweight 25 to <30 kg/m^2: number analyzed (Participants) | 155
    Overweight 25 to <30 kg/m^2 | 46
    Obese >=30 kg/m^2: number analyzed (Participants) | 155
    Obese >=30 kg/m^2 | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Percentage of participants with TEAEs were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial administration of study intervention up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent. TEAEs included both serious and non-serious adverse events.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: Safety analysis set included all participants who received at least 1 dose of esketamine anytime during the 54135419TRD4010 study.
Measure: Number; unit: percentage of participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
percentage of participants | 88.0

2. Primary Outcome: Incidence Rate of Treatment-emergent Adverse Events (TEAEs)
Description: Incidence rate of TEAEs were reported. AE Incidence rate was defined as incidence rate per 100 patient-months = (number of participants with AE divided by sum of days at risk for AE) * 100*365.25/12. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial administration of study intervention up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent. TEAEs included both serious and non-serious adverse events.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: AEs per 100 patient-months
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
AEs per 100 patient-months | 17.33 [14.85 to 20.23]

3. Primary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: Percentage of participants with TESAEs were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial administration of study intervention up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
percentage of participants | 6.0

4. Primary Outcome: Incidence Rate of Treatment-emergent Serious Adverse Events (TESAEs)
Description: Incidence rate of with TESAEs were reported. AE Incidence rate was defined as incidence rate per 100 patient-months = (number of participants with AE divided by sum of days at risk for AE) * 100*365.25/12. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial administration of study intervention up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: AEs per 100 patient-months
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
AEs per 100 patient-months | 0.28 [0.16 to 0.51]

5. Primary Outcome: Percentage of of Participants With TEAEs Leading to Death
Description: Percentage of participants with TEAEs leading to death were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial administration of study intervention up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent. TEAEs included both serious and non-serious adverse events.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
percentage of participants | 0.6 [0.16 to 0.51]

6. Primary Outcome: Incidence Rate of TEAEs Leading to Death
Description: Incidence rate of TEAEs leading to death were reported. AE Incidence rate was defined as incidence rate per 100 patient-months = (number of participants with AE divided by sum of days at risk for AE) * 100*365.25/12. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the intervention. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial administration of study intervention up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent. TEAEs included both serious and non-serious adverse events.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: AEs per 100 patient-months
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
AEs per 100 patient-months | 0.03 [0.00 to 0.18]

7. Primary Outcome: Percentage of Participants With Treatment-emergent AEs of Special Interest (AESIs)
Description: Percentage of participants with TEAEs of special interest were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with intervention. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial administration of study intervention up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent. TEAEs included both serious and non-serious AEs. AEs of special interest were separately grouped by categories sedation, dissociation, suicidality, suggestive of abuse potential, cystitis and hepatic impairment.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
percentage of participants
  Sedation | 16.9
  Dissociation | 12.0
  Suicidality | 3.8
  Suggestive of abuse potential | 37.7
  Cystitis | 0.5

8. Primary Outcome: Incidence Rate of Treatment-emergent AEs of Special Interest (AESIs)
Description: AE Incidence rate: incidence rate per 100 patient-months=(number of participants with AE divided by sum of days at risk for AE)* 100*365.25/12. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with intervention. SAE: AE resulting in any following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Any AE occurring at or after the initial intervention administration up to 30 days after last dose in Study 54135419TRD4010 was considered to be treatment emergent. TEAEs included both serious and non-serious AEs. AEs of special interest were grouped as categories sedation, dissociation, suicidality, suggestive of abuse potential, cystitis and hepatic impairment.
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Population: as for outcome 1
Measure: Number; unit: AEs per 100 patient-months
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
AEs per 100 patient-months
  Sedation | 0.91
  Dissociation | 0.61
  Suicidality | 0.18
  Suggestive of abuse potential | 2.63
  Cystitis | 0.03

9. Primary Outcome: Number of Participants With Suicidal Ideation and Behavior in Study 54135419TRD4010 as Assessed by Columbia-suicide Severity Rating Scale (C-SSRS) Score
Description: Number of participants with suicidal ideation and behavior in study 54135419TRD4010 as assessed by C-SSRS score were reported. C-SSRS score: an assessment tool that evaluated suicidal ideation and behavior. Suicidal ideation (5 items): wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, and active suicidal ideation with specific plan and intent. Suicidal behavior (5 items): preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal), and suicide. Total score from 10 categories was summarized into 3 categories: No suicidal ideation or behavior (0), Suicidal ideation (1 to 5), Suicidal behavior (6 to 10). Total score ranged from 0 to 10. Higher scores indicated more severe suicidal ideation and behavior.
Time Frame: Baseline (Day 1 of Study 54135419TRD3013) up to Week 104 of study 54135419TRD4010 (up to Week 136)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 183
Participants
  No suicidal ideation or behavior | 158
  Suicidal ideation | 24
  Suicidal behavior | 1

10. Secondary Outcome: Percentage of Participants With No Relapse and Without Discontinuation Until the End of the Prospective Observation Period at Week 104
Description: Relapse was defined by any of the following: a) Worsening of depressive symptoms as indicated by Montgomery-Asberg Depression Rating Scale (MADRS) total score >=22 confirmed by 1 additional assessment of MADRS total score >=22 within the next 5 to 31 days. b) Any psychiatric hospitalization for: 1) worsening of depression, 2) suicide prevention or due to a suicide attempt for any of these events. c) Suicide attempt, completed suicide, or any other clinically relevant event determined per investigator's clinical judgment to be indicative of relapse of depressive illness, but for which participant was not hospitalized. MADRS scale consisted of 10 items, scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 0 to 60. Higher scores represented a more severe condition.
Time Frame: Baseline (Day 1 of Study 54135419TRD3013) up to Week 104 of study 54135419TRD4010 (up to Week 136)
Population: Analysis population included participants in remission (MADRS total score of <=10) at any time point during Study 54135419TRD3013.
Measure: Number; unit: percentage of participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 149
percentage of participants | 79.2

11. Secondary Outcome: Change From Baseline of Study 54135419TRD3013 in Clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: Change from baseline of study 54135419TRD3013 in Clinician-rated MADRS total score were reported. MADRS was a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items , scored from 0 (item is not present or normal) to 6 (severe or continuous presence of symptoms), summed up for a total possible score range of 0 to 60. Higher scores represented a more severe condition. The MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts.
Time Frame: Baseline (Day 1 of study 54135419TRD3013) up to weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100, and 104 of study 54135419TRD4010
Population: Efficacy analysis set included all participants who received at least 1 dose of esketamine anytime during the 54135419TRD4010 study. Here, 'N' (Overall number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 181
score on a scale
  Week 4 | -21.9 (8.10)
  Week 8: number analyzed (Participants) | 177
  Week 8 | -21.8 (7.93)
  Week 12: number analyzed (Participants) | 179
  Week 12 | -22.5 (7.25)
  Week 16: number analyzed (Participants) | 175
  Week 16 | -22.8 (7.24)
  Week 20: number analyzed (Participants) | 176
  Week 20 | -22.3 (7.26)
  Week 24: number analyzed (Participants) | 177
  Week 24 | -22.6 (6.82)
  Week 28: number analyzed (Participants) | 173
  Week 28 | -22.4 (7.13)
  Week 32: number analyzed (Participants) | 166
  Week 32 | -22.5 (7.16)
  Week 36: number analyzed (Participants) | 163
  Week 36 | -22.5 (8.12)
  Week 40: number analyzed (Participants) | 163
  Week 40 | -22.7 (7.03)
  Week 44: number analyzed (Participants) | 159
  Week 44 | -22.9 (7.41)
  Week 48: number analyzed (Participants) | 159
  Week 48 | -22.9 (7.19)
  Week 52: number analyzed (Participants) | 151
  Week 52 | -22.6 (7.13)
  Week 56: number analyzed (Participants) | 148
  Week 56 | -23.0 (6.88)
  Week 60: number analyzed (Participants) | 152
  Week 60 | -23.1 (7.11)
  Week 64: number analyzed (Participants) | 151
  Week 64 | -23.4 (7.52)
  Week 68: number analyzed (Participants) | 148
  Week 68 | -23.2 (7.10)
  Week 72: number analyzed (Participants) | 143
  Week 72 | -23.6 (6.98)
  Week 76: number analyzed (Participants) | 138
  Week 76 | -23.8 (6.91)
  Week 80: number analyzed (Participants) | 139
  Week 80 | -23.7 (7.19)
  Week 84: number analyzed (Participants) | 137
  Week 84 | -23.6 (6.87)
  Week 88: number analyzed (Participants) | 134
  Week 88 | -24.4 (6.78)
  Week 92: number analyzed (Participants) | 136
  Week 92 | -24.3 (7.17)
  Week 96: number analyzed (Participants) | 132
  Week 96 | -24.7 (6.57)
  Week 100: number analyzed (Participants) | 130
  Week 100 | -24.9 (6.39)
  Week 104: number analyzed (Participants) | 127
  Week 104 | -25.3 (6.69)

12. Secondary Outcome: Change From Baseline of Study 54135419TRD3013 in Clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS) Score Individual Items
Description: Change from Baseline of Study 54135419TRD3013 in Clinician-rated MADRS Score Individual Items (apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts) were reported. MADRS was a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptoms), summed up for a total possible score range of 0 to 60. Higher scores represent a more severe condition.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 181
score on a scale
  Week 4: Apparent Sadness | -3.0 (1.38)
  Week 8: Apparent Sadness: number analyzed (Participants) | 177
  Week 8: Apparent Sadness | -3.0 (1.45)
  Week 12: Apparent Sadness: number analyzed (Participants) | 179
  Week 12: Apparent Sadness | -3.0 (1.34)
  Week 16: Apparent Sadness: number analyzed (Participants) | 175
  Week 16: Apparent Sadness | -3.1 (1.34)
  Week 20: Apparent Sadness: number analyzed (Participants) | 176
  Week 20: Apparent Sadness | -3.1 (1.31)
  Week 24: Apparent Sadness: number analyzed (Participants) | 177
  Week 24: Apparent Sadness | -2.9 (1.36)
  Week 28: Apparent Sadness: number analyzed (Participants) | 173
  Week 28: Apparent Sadness | -3.0 (1.33)
  Week 32: Apparent Sadness: number analyzed (Participants) | 166
  Week 32: Apparent Sadness | -3.0 (1.28)
  Week 36: Apparent Sadness: number analyzed (Participants) | 163
  Week 36: Apparent Sadness | -3.0 (1.42)
  Week 40: Apparent Sadness: number analyzed (Participants) | 163
  Week 40: Apparent Sadness | -3.0 (1.36)
  Week 44: Apparent Sadness: number analyzed (Participants) | 159
  Week 44: Apparent Sadness | -3.1 (1.38)
  Week 48: Apparent Sadness: number analyzed (Participants) | 159
  Week 48: Apparent Sadness | -3.1 (1.34)
  Week 52: Apparent Sadness: number analyzed (Participants) | 151
  Week 52: Apparent Sadness | -3.1 (1.32)
  Week 56: Apparent Sadness: number analyzed (Participants) | 148
  Week 56: Apparent Sadness | -3.1 (1.23)
  Week 60: Apparent Sadness: number analyzed (Participants) | 152
  Week 60: Apparent Sadness | -3.1 (1.24)
  Week 64: Apparent Sadness: number analyzed (Participants) | 151
  Week 64: Apparent Sadness | -3.2 (1.33)
  Week 68: Apparent Sadness: number analyzed (Participants) | 148
  Week 68: Apparent Sadness | -3.1 (1.23)
  Week 72: Apparent Sadness: number analyzed (Participants) | 143
  Week 72: Apparent Sadness | -3.2 (1.21)
  Week 76: Apparent Sadness: number analyzed (Participants) | 138
  Week 76: Apparent Sadness | -3.3 (1.22)
  Week 80: Apparent Sadness: number analyzed (Participants) | 139
  Week 80: Apparent Sadness | -3.3 (1.24)
  Week 84: Apparent Sadness: number analyzed (Participants) | 137
  Week 84: Apparent Sadness | -3.2 (1.15)
  Week 88: Apparent Sadness: number analyzed (Participants) | 134
  Week 88: Apparent Sadness | -3.4 (1.17)
  Week 92: Apparent Sadness: number analyzed (Participants) | 136
  Week 92: Apparent Sadness | -3.3 (1.20)
  Week 96: Apparent Sadness: number analyzed (Participants) | 132
  Week 96: Apparent Sadness | -3.3 (1.20)
  Week 100: Apparent Sadness: number analyzed (Participants) | 130
  Week 100: Apparent Sadness | -3.4 (1.13)
  Week 104: Apparent Sadness: number analyzed (Participants) | 127
  Week 104: Apparent Sadness | -3.5 (1.20)
  Week 4: Reported Sadness | -3.1 (1.29)
  Week 8: Reported Sadness: number analyzed (Participants) | 177
  Week 8: Reported Sadness | -3.0 (1.38)
  Week 12: Reported Sadness: number analyzed (Participants) | 179
  Week 12: Reported Sadness | -3.0 (1.20)
  Week 16: Reported Sadness: number analyzed (Participants) | 175
  Week 16: Reported Sadness | -3.1 (1.28)
  Week 20: Reported Sadness: number analyzed (Participants) | 176
  Week 20: Reported Sadness | -3.1 (1.24)
  Week 24: Reported Sadness: number analyzed (Participants) | 177
  Week 24: Reported Sadness | -3.1 (1.19)
  Week 28: Reported Sadness: number analyzed (Participants) | 173
  Week 28: Reported Sadness | -3.0 (1.21)
  Week 32: Reported Sadness: number analyzed (Participants) | 166
  Week 32: Reported Sadness | -3.1 (1.18)
  Week 36: Reported Sadness: number analyzed (Participants) | 163
  Week 36: Reported Sadness | -3.0 (1.23)
  Week 40: Reported Sadness: number analyzed (Participants) | 163
  Week 40: Reported Sadness | -3.2 (1.18)
  Week 44: Reported Sadness: number analyzed (Participants) | 159
  Week 44: Reported Sadness | -3.1 (1.23)
  Week 48: Reported Sadness: number analyzed (Participants) | 159
  Week 48: Reported Sadness | -3.1 (1.22)
  Week 52: Reported Sadness: number analyzed (Participants) | 151
  Week 52: Reported Sadness | -3.1 (1.19)
  Week 56: Reported Sadness: number analyzed (Participants) | 148
  Week 56: Reported Sadness | -3.2 (1.12)
  Week 60: Reported Sadness: number analyzed (Participants) | 152
  Week 60: Reported Sadness | -3.3 (1.14)
  Week 64: Reported Sadness: number analyzed (Participants) | 151
  Week 64: Reported Sadness | -3.3 (1.26)
  Week 68: Reported Sadness: number analyzed (Participants) | 148
  Week 68: Reported Sadness | -3.2 (1.24)
  Week 72: Reported Sadness: number analyzed (Participants) | 143
  Week 72: Reported Sadness | -3.2 (1.20)
  Week 76: Reported Sadness: number analyzed (Participants) | 138
  Week 76: Reported Sadness | -3.3 (1.16)
  Week 80: Reported Sadness: number analyzed (Participants) | 139
  Week 80: Reported Sadness | -3.3 (1.12)
  Week 84: Reported Sadness: number analyzed (Participants) | 137
  Week 84: Reported Sadness | -3.3 (1.10)
  Week 88: Reported Sadness: number analyzed (Participants) | 134
  Week 88: Reported Sadness | -3.3 (1.14)
  Week 92: Reported Sadness: number analyzed (Participants) | 136
  Week 92: Reported Sadness | -3.3 (1.24)
  Week 96: Reported Sadness: number analyzed (Participants) | 132
  Week 96: Reported Sadness | -3.4 (1.03)
  Week 100: Reported Sadness: number analyzed (Participants) | 130
  Week 100: Reported Sadness | -3.4 (1.05)
  Week 104: Reported Sadness: number analyzed (Participants) | 127
  Week 104: Reported Sadness | -3.5 (1.07)
  Week 4: Inner Tension | -1.8 (1.19)
  Week 8: Inner Tension: number analyzed (Participants) | 177
  Week 8: Inner Tension | -1.8 (1.18)
  Week 12: Inner Tension: number analyzed (Participants) | 179
  Week 12: Inner Tension | -1.9 (1.20)
  Week 16: Inner Tension: number analyzed (Participants) | 175
  Week 16: Inner Tension | -1.9 (1.15)
  Week 20: Inner Tension: number analyzed (Participants) | 176
  Week 20: Inner Tension | -1.8 (1.19)
  Week 24: Inner Tension: number analyzed (Participants) | 177
  Week 24: Inner Tension | -1.9 (1.21)
  Week 28: Inner Tension: number analyzed (Participants) | 173
  Week 28: Inner Tension | -1.8 (1.23)
  Week 32: Inner Tension: number analyzed (Participants) | 166
  Week 32: Inner Tension | -1.9 (1.23)
  Week 36: Inner Tension: number analyzed (Participants) | 163
  Week 36: Inner Tension | -2.0 (1.07)
  Week 40: Inner Tension: number analyzed (Participants) | 163
  Week 40: Inner Tension | -1.8 (1.17)
  Week 44: Inner Tension: number analyzed (Participants) | 159
  Week 44: Inner Tension | -1.9 (1.20)
  Week 48: Inner Tension: number analyzed (Participants) | 159
  Week 48: Inner Tension | -2.0 (1.25)
  Week 52: Inner Tension: number analyzed (Participants) | 151
  Week 52: Inner Tension | -1.9 (1.16)
  Week 56: Inner Tension: number analyzed (Participants) | 148
  Week 56: Inner Tension | -2.0 (1.20)
  Week 60: Inner Tension: number analyzed (Participants) | 152
  Week 60: Inner Tension | -1.9 (1.32)
  Week 64: Inner Tension: number analyzed (Participants) | 151
  Week 64: Inner Tension | -2.0 (1.34)
  Week 68: Inner Tension: number analyzed (Participants) | 148
  Week 68: Inner Tension | -1.9 (1.26)
  Week 72: Inner Tension: number analyzed (Participants) | 143
  Week 72: Inner Tension | -2.0 (1.26)
  Week 76: Inner Tension: number analyzed (Participants) | 138
  Week 76: Inner Tension | -2.0 (1.22)
  Week 80: Inner Tension: number analyzed (Participants) | 139
  Week 80: Inner Tension | -2.1 (1.13)
  Week 84: Inner Tension: number analyzed (Participants) | 137
  Week 84: Inner Tension | -2.0 (1.28)
  Week 88: Inner Tension: number analyzed (Participants) | 134
  Week 88: Inner Tension | -2.0 (1.20)
  Week 92: Inner Tension: number analyzed (Participants) | 136
  Week 92: Inner Tension | -2.0 (1.16)
  Week 96: Inner Tension: number analyzed (Participants) | 132
  Week 96: Inner Tension | -2.0 (1.14)
  Week 100: Inner Tension: number analyzed (Participants) | 130
  Week 100: Inner Tension | -2.0 (1.18)
  Week 104: Inner Tension: number analyzed (Participants) | 127
  Week 104: Inner Tension | -2.1 (1.22)
  Week 4: Reduced Sleep | -2.1 (1.72)
  Week 8: Reduced Sleep: number analyzed (Participants) | 177
  Week 8: Reduced Sleep | -2.2 (1.64)
  Week 12: Reduced Sleep: number analyzed (Participants) | 179
  Week 12: Reduced Sleep | -2.2 (1.63)
  Week 16: Reduced Sleep: number analyzed (Participants) | 175
  Week 16: Reduced Sleep | -2.2 (1.75)
  Week 20: Reduced Sleep: number analyzed (Participants) | 176
  Week 20: Reduced Sleep | -2.3 (1.72)
  Week 24: Reduced Sleep: number analyzed (Participants) | 177
  Week 24: Reduced Sleep | -2.2 (1.68)
  Week 28: Reduced Sleep: number analyzed (Participants) | 173
  Week 28: Reduced Sleep | -2.2 (1.72)
  Week 32: Reduced Sleep: number analyzed (Participants) | 166
  Week 32: Reduced Sleep | -2.3 (1.70)
  Week 36: Reduced Sleep: number analyzed (Participants) | 163
  Week 36: Reduced Sleep | -2.3 (1.81)
  Week 40: Reduced Sleep: number analyzed (Participants) | 163
  Week 40: Reduced Sleep | -2.3 (1.76)
  Week 44: Reduced Sleep: number analyzed (Participants) | 159
  Week 44: Reduced Sleep | -2.4 (1.61)
  Week 48: Reduced Sleep: number analyzed (Participants) | 159
  Week 48: Reduced Sleep | -2.3 (1.69)
  Week 52: Reduced Sleep: number analyzed (Participants) | 151
  Week 52: Reduced Sleep | -2.2 (1.64)
  Week 56: Reduced Sleep: number analyzed (Participants) | 148
  Week 56: Reduced Sleep | -2.2 (1.73)
  Week 60: Reduced Sleep: number analyzed (Participants) | 152
  Week 60: Reduced Sleep | -2.3 (1.62)
  Week 64: Reduced Sleep: number analyzed (Participants) | 151
  Week 64: Reduced Sleep | -2.2 (1.70)
  Week 68: Reduced Sleep: number analyzed (Participants) | 148
  Week 68: Reduced Sleep | -2.4 (1.82)
  Week 72: Reduced Sleep: number analyzed (Participants) | 143
  Week 72: Reduced Sleep | -2.3 (1.66)
  Week 76: Reduced Sleep: number analyzed (Participants) | 138
  Week 76: Reduced Sleep | -2.4 (1.67)
  Week 80: Reduced Sleep: number analyzed (Participants) | 139
  Week 80: Reduced Sleep | -2.3 (1.84)
  Week 84: Reduced Sleep: number analyzed (Participants) | 137
  Week 84: Reduced Sleep | -2.4 (1.73)
  Week 88: Reduced Sleep: number analyzed (Participants) | 134
  Week 88: Reduced Sleep | -2.5 (1.58)
  Week 92: Reduced Sleep: number analyzed (Participants) | 136
  Week 92: Reduced Sleep | -2.4 (1.70)
  Week 96: Reduced Sleep: number analyzed (Participants) | 132
  Week 96: Reduced Sleep | -2.5 (1.66)
  Week 100: Reduced Sleep: number analyzed (Participants) | 130
  Week 100: Reduced Sleep | -2.5 (1.66)
  Week 104: Reduced Sleep: number analyzed (Participants) | 127
  Week 104: Reduced Sleep | -2.6 (1.76)
  Week 4: Reduced Appetite | -1.7 (1.78)
  Week 8: Reduced Appetite: number analyzed (Participants) | 177
  Week 8: Reduced Appetite | -1.7 (1.75)
  Week 12: Reduced Appetite: number analyzed (Participants) | 179
  Week 12: Reduced Appetite | -1.9 (1.68)
  Week 16: Reduced Appetite: number analyzed (Participants) | 175
  Week 16: Reduced Appetite | -2.0 (1.69)
  Week 20: Reduced Appetite: number analyzed (Participants) | 176
  Week 20: Reduced Appetite | -1.8 (1.74)
  Week 24: Reduced Appetite: number analyzed (Participants) | 177
  Week 24: Reduced Appetite | -1.9 (1.74)
  Week 28: Reduced Appetite: number analyzed (Participants) | 173
  Week 28: Reduced Appetite | -1.9 (1.74)
  Week 32: Reduced Appetite: number analyzed (Participants) | 166
  Week 32: Reduced Appetite | -1.9 (1.72)
  Week 36: Reduced Appetite: number analyzed (Participants) | 163
  Week 36: Reduced Appetite | -1.9 (1.81)
  Week 40: Reduced Appetite: number analyzed (Participants) | 163
  Week 40: Reduced Appetite | -1.9 (1.69)
  Week 44: Reduced Appetite: number analyzed (Participants) | 159
  Week 44: Reduced Appetite | -1.9 (1.81)
  Week 48: Reduced Appetite: number analyzed (Participants) | 159
  Week 48: Reduced Appetite | -1.9 (1.73)
  Week 52: Reduced Appetite: number analyzed (Participants) | 151
  Week 52: Reduced Appetite | -1.9 (1.78)
  Week 56: Reduced Appetite: number analyzed (Participants) | 148
  Week 56: Reduced Appetite | -1.9 (1.65)
  Week 60: Reduced Appetite: number analyzed (Participants) | 152
  Week 60: Reduced Appetite | -1.9 (1.68)
  Week 64: Reduced Appetite: number analyzed (Participants) | 151
  Week 64: Reduced Appetite | -2.0 (1.67)
  Week 68: Reduced Appetite: number analyzed (Participants) | 148
  Week 68: Reduced Appetite | -2.0 (1.69)
  Week 72: Reduced Appetite: number analyzed (Participants) | 143
  Week 72: Reduced Appetite | -2.0 (1.64)
  Week 76: Reduced Appetite: number analyzed (Participants) | 138
  Week 76: Reduced Appetite | -2.0 (1.62)
  Week 80: Reduced Appetite: number analyzed (Participants) | 139
  Week 80: Reduced Appetite | -1.9 (1.78)
  Week 84: Reduced Appetite: number analyzed (Participants) | 137
  Week 84: Reduced Appetite | -2.0 (1.70)
  Week 88: Reduced Appetite: number analyzed (Participants) | 134
  Week 88: Reduced Appetite | -2.0 (1.73)
  Week 92: Reduced Appetite: number analyzed (Participants) | 136
  Week 92: Reduced Appetite | -2.0 (1.67)
  Week 96: Reduced Appetite: number analyzed (Participants) | 132
  Week 96: Reduced Appetite | -2.1 (1.61)
  Week 100: Reduced Appetite: number analyzed (Participants) | 130
  Week 100: Reduced Appetite | -2.0 (1.69)
  Week 104: Reduced Appetite: number analyzed (Participants) | 127
  Week 104: Reduced Appetite | -2.1 (1.72)
  Week 4: Concentration Difficulties | -2.2 (1.28)
  Week 8: Concentration Difficulties: number analyzed (Participants) | 177
  Week 8: Concentration Difficulties | -2.3 (1.37)
  Week 12: Concentration Difficulties: number analyzed (Participants) | 179
  Week 12: Concentration Difficulties | -2.3 (1.26)
  Week 16: Concentration Difficulties: number analyzed (Participants) | 175
  Week 16: Concentration Difficulties | -2.3 (1.28)
  Week 20: Concentration Difficulties: number analyzed (Participants) | 176
  Week 20: Concentration Difficulties | -2.2 (1.25)
  Week 24: Concentration Difficulties: number analyzed (Participants) | 177
  Week 24: Concentration Difficulties | -2.3 (1.26)
  Week 28: Concentration Difficulties: number analyzed (Participants) | 173
  Week 28: Concentration Difficulties | -2.2 (1.28)
  Week 32: Concentration Difficulties: number analyzed (Participants) | 166
  Week 32: Concentration Difficulties | -2.2 (1.23)
  Week 36: Concentration Difficulties: number analyzed (Participants) | 163
  Week 36: Concentration Difficulties | -2.3 (1.28)
  Week 40: Concentration Difficulties: number analyzed (Participants) | 163
  Week 40: Concentration Difficulties | -2.3 (1.21)
  Week 44: Concentration Difficulties: number analyzed (Participants) | 159
  Week 44: Concentration Difficulties | -2.3 (1.26)
  Week 48: Concentration Difficulties: number analyzed (Participants) | 159
  Week 48: Concentration Difficulties | -2.4 (1.18)
  Week 52: Concentration Difficulties: number analyzed (Participants) | 151
  Week 52: Concentration Difficulties | -2.4 (1.20)
  Week 56: Concentration Difficulties: number analyzed (Participants) | 148
  Week 56: Concentration Difficulties | -2.4 (1.14)
  Week 60: Concentration Difficulties: number analyzed (Participants) | 152
  Week 60: Concentration Difficulties | -2.3 (1.19)
  Week 64: Concentration Difficulties: number analyzed (Participants) | 151
  Week 64: Concentration Difficulties | -2.4 (1.25)
  Week 68: Concentration Difficulties: number analyzed (Participants) | 148
  Week 68: Concentration Difficulties | -2.4 (1.26)
  Week 72: Concentration Difficulties: number analyzed (Participants) | 143
  Week 72: Concentration Difficulties | -2.4 (1.10)
  Week 76: Concentration Difficulties: number analyzed (Participants) | 138
  Week 76: Concentration Difficulties | -2.5 (1.17)
  Week 80: Concentration Difficulties: number analyzed (Participants) | 139
  Week 80: Concentration Difficulties | -2.4 (1.10)
  Week 84: Concentration Difficulties: number analyzed (Participants) | 137
  Week 84: Concentration Difficulties | -2.4 (1.14)
  Week 88: Concentration Difficulties: number analyzed (Participants) | 134
  Week 88: Concentration Difficulties | -2.6 (1.08)
  Week 92: Concentration Difficulties: number analyzed (Participants) | 136
  Week 92: Concentration Difficulties | -2.6 (1.12)
  Week 96: Concentration Difficulties: number analyzed (Participants) | 132
  Week 96: Concentration Difficulties | -2.5 (1.10)
  Week 100: Concentration Difficulties: number analyzed (Participants) | 130
  Week 100: Concentration Difficulties | -2.6 (1.06)
  Week 104: Concentration Difficulties: number analyzed (Participants) | 127
  Week 104: Concentration Difficulties | -2.6 (1.10)
  Week 4: Lassitude | -2.5 (1.36)
  Week 8: Lassitude: number analyzed (Participants) | 177
  Week 8: Lassitude | -2.4 (1.33)
  Week 12: Lassitude: number analyzed (Participants) | 179
  Week 12: Lassitude | -2.5 (1.22)
  Week 16: Lassitude: number analyzed (Participants) | 175
  Week 16: Lassitude | -2.5 (1.27)
  Week 20: Lassitude: number analyzed (Participants) | 176
  Week 20: Lassitude | -2.6 (1.33)
  Week 24: Lassitude: number analyzed (Participants) | 177
  Week 24: Lassitude | -2.6 (1.21)
  Week 28: Lassitude: number analyzed (Participants) | 173
  Week 28: Lassitude | -2.6 (1.21)
  Week 32: Lassitude: number analyzed (Participants) | 166
  Week 32: Lassitude | -2.5 (1.20)
  Week 36: Lassitude: number analyzed (Participants) | 163
  Week 36: Lassitude | -2.6 (1.30)
  Week 40: Lassitude: number analyzed (Participants) | 163
  Week 40: Lassitude | -2.5 (1.17)
  Week 44: Lassitude: number analyzed (Participants) | 159
  Week 44: Lassitude | -2.6 (1.16)
  Week 48: Lassitude: number analyzed (Participants) | 159
  Week 48: Lassitude | -2.6 (1.19)
  Week 52: Lassitude: number analyzed (Participants) | 151
  Week 52: Lassitude | -2.6 (1.15)
  Week 56: Lassitude: number analyzed (Participants) | 148
  Week 56: Lassitude | -2.6 (1.16)
  Week 60: Lassitude: number analyzed (Participants) | 152
  Week 60: Lassitude | -2.6 (1.25)
  Week 64: Lassitude: number analyzed (Participants) | 151
  Week 64: Lassitude | -2.6 (1.25)
  Week 68: Lassitude: number analyzed (Participants) | 148
  Week 68: Lassitude | -2.6 (1.21)
  Week 72: Lassitude: number analyzed (Participants) | 143
  Week 72: Lassitude | -2.7 (1.13)
  Week 76: Lassitude: number analyzed (Participants) | 138
  Week 76: Lassitude | -2.6 (1.11)
  Week 80: Lassitude: number analyzed (Participants) | 139
  Week 80: Lassitude | -2.8 (1.00)
  Week 84: Lassitude: number analyzed (Participants) | 137
  Week 84: Lassitude | -2.6 (1.09)
  Week 88: Lassitude: number analyzed (Participants) | 134
  Week 88: Lassitude | -2.8 (1.14)
  Week 92: Lassitude: number analyzed (Participants) | 136
  Week 92: Lassitude | -2.7 (1.09)
  Week 96: Lassitude: number analyzed (Participants) | 132
  Week 96: Lassitude | -2.8 (1.11)
  Week 100: Lassitude: number analyzed (Participants) | 130
  Week 100: Lassitude | -2.9 (1.00)
  Week 104: Lassitude: number analyzed (Participants) | 127
  Week 104: Lassitude | -2.9 (0.91)
  Week 4: Inability to Feel | -2.7 (1.29)
  Week 8: Inability to Feel: number analyzed (Participants) | 177
  Week 8: Inability to Feel | -2.6 (1.34)
  Week 12: Inability to Feel: number analyzed (Participants) | 179
  Week 12: Inability to Feel | -2.7 (1.24)
  Week 16: Inability to Feel: number analyzed (Participants) | 175
  Week 16: Inability to Feel | -2.8 (1.20)
  Week 20: Inability to Feel: number analyzed (Participants) | 176
  Week 20: Inability to Feel | -2.6 (1.19)
  Week 24: Inability to Feel: number analyzed (Participants) | 177
  Week 24: Inability to Feel | -2.8 (1.24)
  Week 28: Inability to Feel: number analyzed (Participants) | 173
  Week 28: Inability to Feel | -2.7 (1.27)
  Week 32: Inability to Feel: number analyzed (Participants) | 166
  Week 32: Inability to Feel | -2.8 (1.30)
  Week 36: Inability to Feel: number analyzed (Participants) | 163
  Week 36: Inability to Feel | -2.8 (1.28)
  Week 40: Inability to Feel: number analyzed (Participants) | 163
  Week 40: Inability to Feel | -2.8 (1.22)
  Week 44: Inability to Feel: number analyzed (Participants) | 159
  Week 44: Inability to Feel | -2.8 (1.26)
  Week 48: Inability to Feel: number analyzed (Participants) | 159
  Week 48: Inability to Feel | -2.7 (1.27)
  Week 52: Inability to Feel: number analyzed (Participants) | 151
  Week 52: Inability to Feel | -2.7 (1.26)
  Week 56: Inability to Feel: number analyzed (Participants) | 148
  Week 56: Inability to Feel | -2.8 (1.22)
  Week 60: Inability to Feel: number analyzed (Participants) | 152
  Week 60: Inability to Feel | -2.9 (1.20)
  Week 64: Inability to Feel: number analyzed (Participants) | 151
  Week 64: Inability to Feel | -2.9 (1.21)
  Week 68: Inability to Feel: number analyzed (Participants) | 148
  Week 68: Inability to Feel | -2.8 (1.14)
  Week 72: Inability to Feel: number analyzed (Participants) | 143
  Week 72: Inability to Feel | -2.8 (1.24)
  Week 76: Inability to Feel: number analyzed (Participants) | 138
  Week 76: Inability to Feel | -2.8 (1.20)
  Week 80: Inability to Feel: number analyzed (Participants) | 139
  Week 80: Inability to Feel | -2.9 (1.29)
  Week 84: Inability to Feel: number analyzed (Participants) | 137
  Week 84: Inability to Feel | -2.9 (1.34)
  Week 88: Inability to Feel: number analyzed (Participants) | 134
  Week 88: Inability to Feel | -2.9 (1.13)
  Week 92: Inability to Feel: number analyzed (Participants) | 136
  Week 92: Inability to Feel | -3.0 (1.20)
  Week 96: Inability to Feel: number analyzed (Participants) | 132
  Week 96: Inability to Feel | -3.0 (1.13)
  Week 100: Inability to Feel: number analyzed (Participants) | 130
  Week 100: Inability to Feel | -3.0 (1.15)
  Week 104: Inability to Feel: number analyzed (Participants) | 127
  Week 104: Inability to Feel | -3.0 (1.23)
  Week 4: Pessimistic Thoughts | -2.0 (1.25)
  Week 8: Pessimistic Thoughts: number analyzed (Participants) | 177
  Week 8: Pessimistic Thoughts | -2.0 (1.24)
  Week 12: Pessimistic Thoughts: number analyzed (Participants) | 179
  Week 12: Pessimistic Thoughts | -2.1 (1.26)
  Week 16: Pessimistic Thoughts: number analyzed (Participants) | 175
  Week 16: Pessimistic Thoughts | -2.1 (1.26)
  Week 20: Pessimistic Thoughts: number analyzed (Participants) | 176
  Week 20: Pessimistic Thoughts | -2.0 (1.25)
  Week 24: Pessimistic Thoughts: number analyzed (Participants) | 177
  Week 24: Pessimistic Thoughts | -2.1 (1.24)
  Week 28: Pessimistic Thoughts: number analyzed (Participants) | 173
  Week 28: Pessimistic Thoughts | -2.1 (1.20)
  Week 32: Pessimistic Thoughts: number analyzed (Participants) | 166
  Week 32: Pessimistic Thoughts | -2.1 (1.23)
  Week 36: Pessimistic Thoughts: number analyzed (Participants) | 163
  Week 36: Pessimistic Thoughts | -2.0 (1.33)
  Week 40: Pessimistic Thoughts: number analyzed (Participants) | 163
  Week 40: Pessimistic Thoughts | -2.1 (1.27)
  Week 44: Pessimistic Thoughts: number analyzed (Participants) | 159
  Week 44: Pessimistic Thoughts | -2.1 (1.23)
  Week 48: Pessimistic Thoughts: number analyzed (Participants) | 159
  Week 48: Pessimistic Thoughts | -2.1 (1.24)
  Week 52: Pessimistic Thoughts: number analyzed (Participants) | 151
  Week 52: Pessimistic Thoughts | -2.0 (1.22)
  Week 56: Pessimistic Thoughts: number analyzed (Participants) | 148
  Week 56: Pessimistic Thoughts | -2.0 (1.25)
  Week 60: Pessimistic Thoughts: number analyzed (Participants) | 152
  Week 60: Pessimistic Thoughts | -2.1 (1.27)
  Week 64: Pessimistic Thoughts: number analyzed (Participants) | 151
  Week 64: Pessimistic Thoughts | -2.1 (1.26)
  Week 68: Pessimistic Thoughts: number analyzed (Participants) | 148
  Week 68: Pessimistic Thoughts | -2.1 (1.21)
  Week 72: Pessimistic Thoughts: number analyzed (Participants) | 143
  Week 72: Pessimistic Thoughts | -2.1 (1.17)
  Week 76: Pessimistic Thoughts: number analyzed (Participants) | 138
  Week 76: Pessimistic Thoughts | -2.1 (1.16)
  Week 80: Pessimistic Thoughts: number analyzed (Participants) | 139
  Week 80: Pessimistic Thoughts | -2.1 (1.23)
  Week 84: Pessimistic Thoughts: number analyzed (Participants) | 137
  Week 84: Pessimistic Thoughts | -2.1 (1.20)
  Week 88: Pessimistic Thoughts: number analyzed (Participants) | 134
  Week 88: Pessimistic Thoughts | -2.1 (1.18)
  Week 92: Pessimistic Thoughts: number analyzed (Participants) | 136
  Week 92: Pessimistic Thoughts | -2.1 (1.21)
  Week 96: Pessimistic Thoughts: number analyzed (Participants) | 132
  Week 96: Pessimistic Thoughts | -2.2 (1.16)
  Week 100: Pessimistic Thoughts: number analyzed (Participants) | 130
  Week 100: Pessimistic Thoughts | -2.2 (1.22)
  Week 104: Pessimistic Thoughts: number analyzed (Participants) | 127
  Week 104: Pessimistic Thoughts | -2.2 (1.18)
  Week 4: Suicidal Thoughts | -0.8 (1.05)
  Week 8: Suicidal Thoughts: number analyzed (Participants) | 177
  Week 8: Suicidal Thoughts | -0.7 (0.97)
  Week 12: Suicidal Thoughts: number analyzed (Participants) | 179
  Week 12: Suicidal Thoughts | -0.8 (1.05)
  Week 16: Suicidal Thoughts: number analyzed (Participants) | 175
  Week 16: Suicidal Thoughts | -0.8 (1.04)
  Week 20: Suicidal Thoughts: number analyzed (Participants) | 176
  Week 20: Suicidal Thoughts | -0.8 (1.01)
  Week 24: Suicidal Thoughts: number analyzed (Participants) | 177
  Week 24: Suicidal Thoughts | -0.8 (1.06)
  Week 28: Suicidal Thoughts: number analyzed (Participants) | 173
  Week 28: Suicidal Thoughts | -0.8 (1.02)
  Week 32: Suicidal Thoughts: number analyzed (Participants) | 166
  Week 32: Suicidal Thoughts | -0.8 (1.01)
  Week 36: Suicidal Thoughts: number analyzed (Participants) | 163
  Week 36: Suicidal Thoughts | -0.7 (1.13)
  Week 40: Suicidal Thoughts: number analyzed (Participants) | 163
  Week 40: Suicidal Thoughts | -0.8 (0.97)
  Week 44: Suicidal Thoughts: number analyzed (Participants) | 159
  Week 44: Suicidal Thoughts | -0.7 (0.91)
  Week 48: Suicidal Thoughts: number analyzed (Participants) | 159
  Week 48: Suicidal Thoughts | -0.8 (0.98)
  Week 52: Suicidal Thoughts: number analyzed (Participants) | 151
  Week 52: Suicidal Thoughts | -0.8 (0.98)
  Week 56: Suicidal Thoughts: number analyzed (Participants) | 148
  Week 56: Suicidal Thoughts | -0.8 (0.99)
  Week 60: Suicidal Thoughts: number analyzed (Participants) | 152
  Week 60: Suicidal Thoughts | -0.8 (0.97)
  Week 64: Suicidal Thoughts: number analyzed (Participants) | 151
  Week 64: Suicidal Thoughts | -0.8 (0.98)
  Week 68: Suicidal Thoughts: number analyzed (Participants) | 148
  Week 68: Suicidal Thoughts | -0.8 (0.98)
  Week 72: Suicidal Thoughts: number analyzed (Participants) | 143
  Week 72: Suicidal Thoughts | -0.8 (1.01)
  Week 76: Suicidal Thoughts: number analyzed (Participants) | 138
  Week 76: Suicidal Thoughts | -0.8 (1.01)
  Week 80: Suicidal Thoughts: number analyzed (Participants) | 139
  Week 80: Suicidal Thoughts | -0.8 (1.03)
  Week 84: Suicidal Thoughts: number analyzed (Participants) | 137
  Week 84: Suicidal Thoughts | -0.8 (0.97)
  Week 88: Suicidal Thoughts: number analyzed (Participants) | 134
  Week 88: Suicidal Thoughts | -0.8 (0.98)
  Week 92: Suicidal Thoughts: number analyzed (Participants) | 136
  Week 92: Suicidal Thoughts | -0.8 (0.97)
  Week 96: Suicidal Thoughts: number analyzed (Participants) | 132
  Week 96: Suicidal Thoughts | -0.8 (1.04)
  Week 100: Suicidal Thoughts: number analyzed (Participants) | 130
  Week 100: Suicidal Thoughts | -0.8 (1.03)
  Week 104: Suicidal Thoughts: number analyzed (Participants) | 127
  Week 104: Suicidal Thoughts | -0.8 (1.01)

13. Secondary Outcome: Change From Baseline of Study 54135419TRD3013 in Clinical Global Impression -Severity (CGI-S) Scale Score
Description: Change from Baseline of Study 54135419TRD3013 in CGI-S scale score were reported. The CGI-S provided an overall clinician-determined summary measure of the severity of the participant's illness that took into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluated the severity of psychopathology on a scale of 1 to 7: where, 1 = normal (not ill); 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participant's. Negative change in score indicated improvement. Participant's with a score of zero were considered missing.
Time Frame: as for outcome 11
Population: Efficacy analysis set included all subjects who received at least 1 dose of esketamine anytime during the 54135419TRD4010 study. Here, 'N' (Overall number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 181
score on a scale
  Week 4 | -2.5 (1.00)
  Week 8: number analyzed (Participants) | 177
  Week 8 | -2.6 (1.02)
  Week 12: number analyzed (Participants) | 179
  Week 12 | -2.6 (0.99)
  Week 16: number analyzed (Participants) | 175
  Week 16 | -2.6 (0.96)
  Week 20: number analyzed (Participants) | 176
  Week 20 | -2.6 (0.96)
  Week 24: number analyzed (Participants) | 174
  Week 24 | -2.7 (0.96)
  Week 28: number analyzed (Participants) | 172
  Week 28 | -2.8 (0.96)
  Week 32: number analyzed (Participants) | 166
  Week 32 | -2.7 (1.01)
  Week 36: number analyzed (Participants) | 162
  Week 36 | -2.7 (0.99)
  Week 40: number analyzed (Participants) | 162
  Week 40 | -2.9 (0.99)
  Week 44: number analyzed (Participants) | 159
  Week 44 | -2.9 (0.98)
  Week 48: number analyzed (Participants) | 158
  Week 48 | -2.9 (0.96)
  Week 52: number analyzed (Participants) | 151
  Week 52 | -2.8 (1.00)
  Week 56: number analyzed (Participants) | 148
  Week 56 | -2.9 (0.93)
  Week 60: number analyzed (Participants) | 152
  Week 60 | -2.9 (0.96)
  Week 64: number analyzed (Participants) | 150
  Week 64 | -2.9 (0.99)
  Week 68: number analyzed (Participants) | 146
  Week 68 | -2.9 (0.93)
  Week 72: number analyzed (Participants) | 142
  Week 72 | -2.9 (0.93)
  Week 76: number analyzed (Participants) | 138
  Week 76 | -2.9 (0.93)
  Week 80: number analyzed (Participants) | 139
  Week 80 | -2.9 (0.91)
  Week 84: number analyzed (Participants) | 137
  Week 84 | -3.0 (0.86)
  Week 88: number analyzed (Participants) | 133
  Week 88 | -3.0 (0.88)
  Week 92: number analyzed (Participants) | 135
  Week 92 | -3.0 (0.88)
  Week 96: number analyzed (Participants) | 132
  Week 96 | -3.1 (0.88)
  Week 100: number analyzed (Participants) | 130
  Week 100 | -3.1 (0.87)
  Week 104: number analyzed (Participants) | 123
  Week 104 | -3.1 (0.85)

14. Secondary Outcome: Change From Baseline of Study 54135419TRD3013 in Patient Health Questionnaire (PHQ) 9-item Total Score
Description: Change from Baseline of Study 54135419TRD3013 in PHQ 9-item total score were reported. The PHQ-9 was a validated 9-item, patient-reported outcome (PRO) measure to assess depressive symptoms. Each item was rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses were summed to a total score with a range of 0 to 27. Higher scores indicated greater severity of depressive symptoms.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 178
score on a scale
  Week 4 | -11.0 (5.80)
  Week 8: number analyzed (Participants) | 174
  Week 8 | -10.9 (5.98)
  Week 12: number analyzed (Participants) | 175
  Week 12 | -10.9 (5.73)
  Week 16: number analyzed (Participants) | 173
  Week 16 | -11.2 (5.53)
  Week 20: number analyzed (Participants) | 171
  Week 20 | -11.3 (5.46)
  Week 24: number analyzed (Participants) | 173
  Week 24 | -11.3 (5.19)
  Week 28: number analyzed (Participants) | 172
  Week 28 | -11.5 (5.25)
  Week 32: number analyzed (Participants) | 161
  Week 32 | -11.3 (5.71)
  Week 36: number analyzed (Participants) | 158
  Week 36 | -11.6 (6.06)
  Week 40: number analyzed (Participants) | 159
  Week 40 | -11.5 (5.55)
  Week 44: number analyzed (Participants) | 155
  Week 44 | -11.9 (5.67)
  Week 48: number analyzed (Participants) | 156
  Week 48 | -11.9 (5.61)
  Week 52: number analyzed (Participants) | 149
  Week 52 | -11.4 (5.55)
  Week 56: number analyzed (Participants) | 145
  Week 56 | -12.0 (5.19)
  Week 60: number analyzed (Participants) | 150
  Week 60 | -11.9 (5.24)
  Week 64: number analyzed (Participants) | 148
  Week 64 | -11.9 (5.18)
  Week 68: number analyzed (Participants) | 145
  Week 68 | -11.9 (5.60)
  Week 72: number analyzed (Participants) | 139
  Week 72 | -12.1 (5.00)
  Week 76: number analyzed (Participants) | 135
  Week 76 | -12.2 (5.12)
  Week 80: number analyzed (Participants) | 134
  Week 80 | -12.1 (5.28)
  Week 84: number analyzed (Participants) | 134
  Week 84 | -11.9 (5.19)
  Week 88: number analyzed (Participants) | 129
  Week 88 | -12.2 (5.21)
  Week 92: number analyzed (Participants) | 133
  Week 92 | -12.5 (5.11)
  Week 96: number analyzed (Participants) | 129
  Week 96 | -12.2 (5.10)
  Week 100: number analyzed (Participants) | 127
  Week 100 | -12.7 (4.78)
  Week 104: number analyzed (Participants) | 125
  Week 104 | -12.7 (4.97)

15. Secondary Outcome: Change From Baseline of Study 54135419TRD3013 in European Quality of Life (EuroQol) 5 Dimension 5-Level (EQ-5D-5L): Health Status Index
Description: Change from baseline of Study 54135419TRD3013 in EQ-5D-5LQuestionnaire Score: health status index were reported. The EQ-5D-5L descriptive system comprised the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions were divided into 5 levels of perceived problems (level 1 = no problem, level 2 = slight problems, level 3 = moderate problems, level 4 = severe problems, level 5 = extreme problems). The participant selected an answer for each of the 5 dimensions considering a response that best matched participant's health "today." Responses were used to generate health status index ranged from -0.594 to 1 (where 1 represents full health and negative values represent health states considered worse than dead). Positive change in score indicated improvement.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 178
score on a scale
  Week 4: number analyzed (Participants) | 177
  Week 4 | 0.323 (0.2479)
  Week 8: number analyzed (Participants) | 173
  Week 8 | 0.320 (0.2518)
  Week 12 | 0.325 (0.2379)
  Week 16: number analyzed (Participants) | 172
  Week 16 | 0.322 (0.2568)
  Week 20: number analyzed (Participants) | 175
  Week 20 | 0.336 (0.2444)
  Week 24: number analyzed (Participants) | 175
  Week 24 | 0.331 (0.2337)
  Week 28: number analyzed (Participants) | 171
  Week 28 | 0.323 (0.2415)
  Week 32: number analyzed (Participants) | 163
  Week 32 | 0.335 (0.2377)
  Week 36: number analyzed (Participants) | 160
  Week 36 | 0.341 (0.2512)
  Week 40: number analyzed (Participants) | 161
  Week 40 | 0.333 (0.2364)
  Week 44: number analyzed (Participants) | 157
  Week 44 | 0.343 (0.2576)
  Week 48: number analyzed (Participants) | 158
  Week 48 | 0.345 (0.2317)
  Week 52: number analyzed (Participants) | 150
  Week 52 | 0.332 (0.2374)
  Week 56: number analyzed (Participants) | 146
  Week 56 | 0.348 (0.2348)
  Week 60: number analyzed (Participants) | 150
  Week 60 | 0.364 (0.2322)
  Week 64: number analyzed (Participants) | 150
  Week 64 | 0.350 (0.2422)
  Week 68: number analyzed (Participants) | 146
  Week 68 | 0.337 (0.2546)
  Week 72: number analyzed (Participants) | 142
  Week 72 | 0.354 (0.2295)
  Week 76: number analyzed (Participants) | 135
  Week 76 | 0.357 (0.2440)
  Week 80: number analyzed (Participants) | 138
  Week 80 | 0.362 (0.2375)
  Week 84: number analyzed (Participants) | 134
  Week 84 | 0.350 (0.2295)
  Week 88: number analyzed (Participants) | 133
  Week 88 | 0.366 (0.2385)
  Week 92: number analyzed (Participants) | 134
  Week 92 | 0.367 (0.2275)
  Week 96: number analyzed (Participants) | 130
  Week 96 | 0.375 (0.2333)
  Week 100: number analyzed (Participants) | 129
  Week 100 | 0.387 (0.2321)
  Week 104: number analyzed (Participants) | 125
  Week 104 | 0.387 (0.2444)

16. Secondary Outcome: Change From Baseline of Study 54135419TRD3013 in European Quality of Life (EuroQol) 5 Dimension 5-Level (EQ-5D-5L): Visual Analogue Scale (VAS)
Description: Change from baseline of Study 54135419TRD3013 in EQ-5D-5L: visual analogue scale were reported. EQ-VAS self-rating recorded the participant's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicated improvement.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD)
Number analyzed (Participants) | 175
score on a scale
  Week 4: number analyzed (Participants) | 174
  Week 4 | 27.35 (20.595)
  Week 8: number analyzed (Participants) | 174
  Week 8 | 26.24 (21.939)
  Week 12 | 26.74 (20.884)
  Week 16: number analyzed (Participants) | 173
  Week 16 | 27.98 (20.523)
  Week 20: number analyzed (Participants) | 174
  Week 20 | 27.85 (20.143)
  Week 24: number analyzed (Participants) | 174
  Week 24 | 28.83 (20.438)
  Week 28: number analyzed (Participants) | 172
  Week 28 | 28.23 (21.006)
  Week 32: number analyzed (Participants) | 162
  Week 32 | 28.30 (21.119)
  Week 36: number analyzed (Participants) | 159
  Week 36 | 29.99 (19.901)
  Week 40: number analyzed (Participants) | 160
  Week 40 | 28.56 (21.210)
  Week 44: number analyzed (Participants) | 156
  Week 44 | 29.19 (21.259)
  Week 48: number analyzed (Participants) | 156
  Week 48 | 29.57 (21.717)
  Week 52: number analyzed (Participants) | 149
  Week 52 | 29.60 (21.419)
  Week 56: number analyzed (Participants) | 145
  Week 56 | 29.90 (20.828)
  Week 60: number analyzed (Participants) | 150
  Week 60 | 30.47 (20.423)
  Week 64: number analyzed (Participants) | 149
  Week 64 | 30.49 (20.352)
  Week 68: number analyzed (Participants) | 146
  Week 68 | 29.82 (20.195)
  Week 72: number analyzed (Participants) | 141
  Week 72 | 30.84 (20.252)
  Week 76: number analyzed (Participants) | 134
  Week 76 | 31.90 (19.866)
  Week 80: number analyzed (Participants) | 137
  Week 80 | 31.23 (20.512)
  Week 84: number analyzed (Participants) | 133
  Week 84 | 30.40 (19.697)
  Week 88: number analyzed (Participants) | 132
  Week 88 | 31.10 (20.469)
  Week 92: number analyzed (Participants) | 133
  Week 92 | 31.87 (20.228)
  Week 96: number analyzed (Participants) | 130
  Week 96 | 30.75 (19.759)
  Week 100: number analyzed (Participants) | 128
  Week 100 | 31.66 (18.887)
  Week 104: number analyzed (Participants) | 125
  Week 104 | 33.75 (19.356)

ADVERSE EVENTS:
Time Frame: From Day 1 of study 54135419TRD4010 up to 30 days after last dose of study drug at Week 104 (up to Week 108)
Description: Safety analysis set included all participants who received at least 1 dose of esketamine anytime during the 54135419TRD4010 study.
Groups:
- Esketamine + Oral AD: Participants (who received esketamine nasal spray in study 54135419TRD3013 [NCT04338321] through Week 30 [every 2 weeks dosing] or Week 31 [once weekly dosing],and completed the maintenance phase at Week 32), received flexible dose of esketamine nasal spray 28 milligrams (mg) (one spray to each nostril at 0 minute), 56 mg (one spray to each nostril at 0 and 5 minutes) or 84 mg (one spray to each nostril at 0, 5 and 105 minutes) once weekly or every 2 weeks from Day 1 (Week 32 visit of study 54135419TRD3013 until week 104 along with oral AD, serotonin-norepinephrine reuptake inhibitor/selective serotonin reuptake inhibitor (SSRI/SNRI) in this long-term extension (LTE) study. Time 0 minute signified time of first esketamine nasal spray administration to 1 nostril. Esketamine nasal devices contained a total of 28 mg esketamine per device (2 sprays). Only one device was used at a timepoint.
Arm/Group | Esketamine + Oral AD
All-Cause Mortality (participants affected / at risk) | 1/183
Serious Adverse Events (participants affected / at risk) | 11/183
Other Adverse Events (participants affected / at risk) | 145/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esketamine + Oral AD (N=183)
Acute coronary syndrome (Cardiac disorders) | 1
Goitre (Endocrine disorders) | 1
Macular hole (Eye disorders) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esketamine + Oral AD (N=183)
Vertigo (Ear and labyrinth disorders) | 32
Lacrimation increased (Eye disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 37
Vomiting (Gastrointestinal disorders) | 12
COVID-19 (Infections and infestations) | 30
Nasopharyngitis (Infections and infestations) | 37
Blood pressure increased (Investigations) | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 20
Dizziness (Nervous system disorders) | 50
Dysgeusia (Nervous system disorders) | 14
Headache (Nervous system disorders) | 81
Paraesthesia (Nervous system disorders) | 13
Somnolence (Nervous system disorders) | 24
Dissociation (Psychiatric disorders) | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13
Sneezing (Respiratory, thoracic and mediastinal disorders) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/18/NCT04829318/Prot_002.pdf
  • Statistical Analysis Plan (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT04829318/SAP_003.pdf